CLINICAL TRIAL: NCT03079414
Title: The Role of Electrophysiology Testing in Survivors of Unexplained Cardiac Arrest
Acronym: EPS ARREST
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 108939
Record Dates: First submitted 2017-03-02; First posted 2017-03-14 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Sudden Cardiac Death
Keywords: Sudden Cardiac Death; Cardiac Arrhythmia; Electrophysiology Study; Genetics
MeSH Terms: conditions — Death, Sudden, Cardiac; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will attempted to be collected for all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Unexplained Aborted Cardiac Arrest: Survivors of sudden cardiac death with no identifiable etiology following initial diagnostic workup.
  Interventions: Procedure: Invasive Electrophysiology Study

INTERVENTIONS:
Procedure: Invasive Electrophysiology Study — Invasive electrophysiology studies will be performed using four catheters placed in the right ventricular apex, the coronary sinus, the His bundle region, and the high right atrium. Standard induction protocols for supraventricular and ventricular arrhythmias will be utilized in the absence and presence of isoproterenol. Long-short ventricular extra-stimuli will also be delivered to screen for bundle branch reentrant ventricular tachycardia. The study is considered observational as the participating sites perform electrophysiology studies in this patient population as part of standard clinical care.

SUMMARY:
Sudden cardiac death (SCD) remains a major cause of mortality within developed nations despite aggressive efforts to reduce its societal burden. Despite extensive clinical and genetic investigations, a subgroup of cardiac arrests remain unexplained, highlighting the potential contribution of additional cardiac conditions that may not be identified with contemporary diagnostic algorithms. The EPS ARREST study aims to evaluate the role of invasive electrophysiology study within this patient population.

DETAILED DESCRIPTION:
The majority of cases of SCD in older individuals occur secondary to coronary and structural heart disease, while genetic channelopathies and cardiomyopathies are prominent contributors in young adults. Among individuals that suffer aborted cardiac arrests in the absence of overt coronary and structural heart disease, diagnostic algorithms that screen for cardiac channelopathies and more subtle forms of structural heart disease have been established. Despite the extensive investigations currently utilized, a significant proportion of aborted cardiac arrests remain unexplained.

Although invasive electrophysiology studies are a cornerstone for diagnosis and management of arrhythmia disorders, they are not invariably included in the workup of cases of unexplained aborted cardiac arrest. This is largely driven by initial studies suggesting that the diagnostic yield in this context is low, however these investigations often used invasive electrophysiology studies indiscriminately in all cases of aborted cardiac arrest. Since these earlier studies, our insight and approach to SCD has evolved and it has become clear that the majority of patients do not require an invasive electrophysiology study for diagnosis. However an invasive electrophysiology study may still have an important role among these individuals when the initial workup is negative. Notably, arrhythmias that require invasive electrophysiology for diagnosis, including bundle branch reentrant ventricular tachycardia and supraventricular tachycardias associated with hemodynamic collapse, have been identified as arrhythmic culprits in this patient population.

The goal of the EPS ARREST study is to evaluate the diagnostic yield of a standardized invasive electrophysiology study among survivors of SCD when initial investigations fail to identify an underlying etiology.

ELIGIBILITY:
Inclusion Criteria:

1. Unexplained cardiac arrest requiring cardioversion or defibrillation
2. Willing and able to sign informed consent

Exclusion Criteria:

1. Coronary artery disease (stenosis > 50%) and clinical findings consistent with an ischemic arrest
2. Reduced left ventricular function (left ventricular ejection fraction < 50%) on echocardiogram or cardiac MRI.
3. Persistent resting QTc > 460 msec for males and 480 msec for females
4. Resting QTc < 350 msec
5. Type I Brugada ECG with >/= 2 mm ST elevation in V1 and/or V2 (Spontaneous or Drug-Induced)
6. Polymorphic or bidirectional ventricular tachycardia observed with exertion on exercise treadmill testing
7. Clinical, electrocardiographic, and/or imaging findings consistent with a diagnosis of arrhythmogenic right ventricular cardiomyopathy
8. Myocarditis
9. Reversible cause of cardiac arrest such as marked hypokalemia (<2.8 mmol/l) or drug overdose sufficient in severity without other cause to explain the cardiac arrest.
10. Arrhythmic mitral valve prolapse syndrome
11. Documented ventricular fibrillation initiated by a short-coupled premature ventricular contraction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Survivors of unexplained sudden cardiac death for whom an underlying etiology remains unclear following a standard diagnostic workup, including 12-lead surface ECG, coronary artery assessment, echocardiography, cardiac MRI with late gadolinium enhancement, procainamide challenge, and exercise treadmill testing.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Arrhythmic culprit for aborted cardiac arrest | Assessed immediately upon testing
  Identification of an arrhythmic culprit for aborted cardiac arrest using an invasive electrophysiology study.

SECONDARY OUTCOMES:
Prevalence of bundle branch reentrant ventricular tachycardia | Assessed immediately upon testing
  Prevalence of bundle branch reentrant ventricular tachycardia among survivors of unexplained cardiac arrest.
Prevalence of supraventricular tachycardia associated with hemodynamic collapse | Assessed immediately upon testing
  Prevalence of inducible supraventricular tachycardia during invasive electrophysiology study among survivors of unexplained cardiac arrest.
Prevalence of a latent/cryptic accessory pathway | Assessed immediately upon testing.
  Prevalence of a latent/cryptic accessory pathway among survivors of unexplained cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Roberts, MD MAS, Principal Investigator — Western University; Andrew D Krahn, MD, Study Director — University of British Columbia; Melvin M Scheinman, MD, Study Director — University of California, San Francisco
Locations (21):
- United States (11):
  - UCLA Medical Center, Los Angeles, California
  - UC San Diego Health System, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - Queen's Medical Center, Honolulu, Hawaii
  - Massachusetts General Hospital, Boston, Massachusetts
  - Regions Hospital, Saint Paul, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Laval University, Québec, Quebec
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD with other researchers.

REFERENCES:
- [Background] Krahn AD, Healey JS, Chauhan V, Birnie DH, Simpson CS, Champagne J, Gardner M, Sanatani S, Exner DV, Klein GJ, Yee R, Skanes AC, Gula LJ, Gollob MH. Systematic assessment of patients with unexplained cardiac arrest: Cardiac Arrest Survivors With Preserved Ejection Fraction Registry (CASPER). Circulation. 2009 Jul 28;120(4):278-85. doi: 10.1161/CIRCULATIONAHA.109.853143. Epub 2009 Jul 13. PMID 19597050
- [Background] Wang YS, Scheinman MM, Chien WW, Cohen TJ, Lesh MD, Griffin JC. Patients with supraventricular tachycardia presenting with aborted sudden death: incidence, mechanism and long-term follow-up. J Am Coll Cardiol. 1991 Dec;18(7):1711-9. doi: 10.1016/0735-1097(91)90508-7. PMID 1960318
- [Background] Roberts JD, Gollob MH, Young C, Connors SP, Gray C, Wilton SB, Green MS, Zhu DW, Hodgkinson KA, Poon A, Li Q, Orr N, Tang AS, Klein GJ, Wojciak J, Campagna J, Olgin JE, Badhwar N, Vedantham V, Marcus GM, Kwok PY, Deo RC, Scheinman MM. Bundle Branch Re-Entrant Ventricular Tachycardia: Novel Genetic Mechanisms in a Life-Threatening Arrhythmia. JACC Clin Electrophysiol. 2017 Mar;3(3):276-288. doi: 10.1016/j.jacep.2016.09.019. Epub 2016 Dec 21. PMID 29759522